CLINICAL TRIAL: NCT01649856
Title: A Comparative, Randomized, Parallel-group, Multi-center, Phase IIIB Study to Investigate the Efficacy of Subcutaneous (SC) Rituximab Versus Intravenous (IV) Rituximab Both in Combination With CHOP (R-CHOP) in Previously Untreated Patients With CD20-positive Diffuse Large B-cell Lymphoma (DLBCL)
Brief Title: A Study of Subcutaneous Versus Intravenous MabThera/Rituxan (Rituximab) in Combination With CHOP Chemotherapy in Patients With Previously Untreated CD20-Positive Diffuse Large B-Cell Lymphoma
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MO28107; 2012-000669-19 (EudraCT Number)
Record Dates: First submitted 2012-07-23; First posted 2012-07-25 (Estimated); Results first posted 2016-02-12 (Estimated); Last update posted 2017-10-11 (Actual); Status verified 2017-09

CONDITIONS: Lymphoma, Large B-Cell, Diffuse
MeSH Terms: conditions — Lymphoma, Large B-Cell, Diffuse | interventions — Rituximab

ARMS (2):
- A: Rituximab SC (Experimental)
  Interventions: Drug: CHOP; Drug: rituximab [MabThera/Rituxan]
- B: Rituximab IV (Active Comparator)
  Interventions: Drug: CHOP; Drug: rituximab [MabThera/Rituxan]

INTERVENTIONS:
Drug: CHOP — CHOP chemotherapy: cyclophosphamide, doxorubicin, vincristine, prednisone/prednisolone; 6 or 8 cycles
Drug: rituximab [MabThera/Rituxan] — The first rituximab dose will be administered intravenously on Day of Cycle 1 at a dose of 375 mg/m2. Subsequent doses of 1400 mg are administered subcutaneously on Day 1 of each cycle, for a further 7 cycles
  Arms: A: Rituximab SC
Drug: rituximab [MabThera/Rituxan] — 375 mg/m2 intravenously on Day 1 of each cycle, 8 cycles
  Arms: B: Rituximab IV

SUMMARY:
This multicenter, randomized, open label parallel-group study will evaluate the efficacy and safety of subcutaneous versus intravenous MabThera/Rituxan (rituximab) in combination with CHOP chemotherapy in patients with previously untreated CD20-positive diffuse large B-Cell lymphoma. Patients will be randomized to receive either MabThera/Rituxan 1400 mg subcutaneously or MabThera/Rituxan 375 mg/m2 intravenously on Day 1 of each cycle for 8 cycles, in combination with 6-8 cycles of CHOP chemotherapy. Anticipated time on study treatment is 6 months.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients, >/= 18 and </= 80 years of age at time of study inclusion
* Histologically confirmed, previously untreated CD20-positive diffuse large B-cell lymphoma (DLBCL) according to the WHO classification system
* Patients with an International Prognostic Index (IPI) score 1-5, or IPI score 0 with bulky disease, defined as one lesion >/= 7.5 cm
* At least one bi-dimensionally measurable lesion defined as >/= 1.5 cm in its largest dimension on CT scan, PET-CT scan or MRI
* Adequate hematologic function
* Eastern Cooperative Oncology Group (EOCD) performance status </= 2

Exclusion Criteria:

* Primary or secondary central nervous system lymphoma, histologic evidence of transformation to Burkitt lymphoma, primary mediastinal DLBCL, primary effusion lymphoma, primary cutaneous DLBCL, or primary DLBCL of the testis
* Transformed lymphoma or follicular lymphoma IIIB
* Prior therapy for DLBCL, with the exception of nodal biopsy or local irradiation
* History of other malignancy, except for curatively treated basal or squamous cell carcinoma or melanoma of the skin, carcinoma in situ of the cervix, or a malignancy that has been treated without curative intent and has been in remission without treatment for >/= 5 years prior to enrolment
* Inadequate renal or hepatic function
* Known human immunodeficiency virus (HIV) infection or HIV seropositive status
* Active hepatitis B virus (HBV) or active hepatitis C virus (HCV) infection. Patients with occult or prior HBV infection as defined by protocol may be included. Patients positive for HCV antibody are eligible only if polymerase chain reaction testing for HCV ribonucleic acid is negative.
* History of severe allergic or anaphylactic reactions to humanized or murine monoclonal antibodies or known sensitivity or allergy to murine products
* Contraindication to any of the individual components of CHOP, including prior receipt of anthracyclines
* Prior treatment with cytotoxic drugs or rituximab for another condition (e.g. rheumatoid arthritis) or prior use of an anti-CD20 antibody
* Pregnant or lactating women

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 572 (Actual)
Dates: Start 2012-08-24 (Actual); Primary Completion 2014-10-21 (Actual); Study Completion 2016-09-16 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (186):
- Algeria (2):
  - EHS CAC Hospital FRANTZ FANON ZABANA BLIDA; Hematology ward, Blida
  - Centre hospitalo-univerisitaire de Tizi Ouzou - Nedir Mohamed;Service d'hématologie, Tizi Ouzou
- Argentina (2):
  - Cemic; Haematology, Buenos Aires
  - Hospital Privado de Comunidad; Oncology, Mar del Plata
- Belgium (11):
  - Onze Lieve Vrouwziekenhuis Aalst, Aalst
  - ZNA Middelheim, Antwerp
  - CHU Brugmann (Victor Horta), Brussels
  - Clin Univ de Bxl Hôpital Erasme, Brussels
  - CHU Charleroi-ISPPC-Espace Santé, Charleroi
  - CHU de Charleroi, Charleroi
  - GHdC Site Notre Dame, Charleroi
  - UZ Gent, Ghent
  - Jessa Zkh (Campus Virga Jesse), Hasselt
  - AZ Turnhout Sint Elisabeth, Turnhout
  - CHR de Verviers - East Belgium, Verviers
- Brazil (6):
  - Crio - Centro Regional Integrado de Oncologia, Fortaleza, Ceará
  - Instituto Nacional de Cancer - INCa; Oncologia, Rio de Janeiro, Rio de Janeiro
  - Clinicas Oncologicas Integradas - COI, Rio de Janeiro, Rio de Janeiro
  - Hospital Giovanni Battista - Mae de Deus Center; Instituto do Cancer, Porto Alegre, Rio Grande do Sul
  - Hospital Amaral Carvalho, Jaú, São Paulo
  - Hospital das Clinicas - FMUSP; Hematologia, São Paulo, São Paulo
- Bulgaria (3):
  - University Hospital Sv.Georgi Clnic of Hematology; Hematology, Plovdiv
  - Military Medical Academy; Hematology And Oncology, Sofia
  - UMHAT Alexandrovska EAD; Hematology, Sofia
- Canada (10):
  - Lion'S Gate Hospital, North Vancouver, British Columbia
  - Cancer Care Manitoba, Winnipeg, Manitoba
  - Regional health authority A vitalite health network, Moncton, New Brunswick
  - Royal Victoria Regional Health Centre; c/o Oncology Clinical Trials, Barrie, Ontario
  - William Osler Health System Brampton Civic Hospital, Brampton, Ontario
  - Grand River Regional Cancer Centre, Kitchener, Ontario
  - Southlake Regional Health Center; Community Care Clinic / Oncology, Newmarket, Ontario
  - Toronto East General Hospital; Haematology/Oncology, Toronto, Ontario
  - University Health Network; Princess Margaret Hospital; Medical Oncology Dept, Toronto, Ontario
  - Windsor Regional Cancer Centre, Windsor, Ontario
- Colombia (2):
  - Clínica Imbanaco; Oncology, Cali
  - Hospital Pablo Tobon Uribe, Medellin-Antioquia
- Finland (5):
  - Helsinki University Central Hospital; Dept of Oncology, Helsinki
  - Middle Finland Central Hospital, Jyväskylä
  - Oulu University Hospital; Oncology, Oulu
  - Tampere University Hospital; Dept of Oncology, Tampere
  - Turku Uni Central Hospital; Oncology Clinics, Turku
- France (10):
  - Ch Victor Dupouy; Hematologie, Argenteuil
  - Hopital Augustin Morvan; Hematologie, Brest
  - Ch Du Mans; Medecine Hematologie Oncologie, Le Mans
  - Centre ONCOGARD - Institut de Cancerologie du Gard, Nîmes
  - Hopital Yves Le Foll; Hematologie Oncologie, Saint-Brieuc
  - Ch De Saint Quentin; Medecine B10, Saint-Quentin
  - Hopital Sud; Hematologie Clinique, Salouël
  - Clinique Ste Anne, Strasbourg
  - Hopital Hautepierre; Hematologie Oncologie, Strasbourg
  - Hia Sainte Anne; Medecine Interne Oncologie, Toulon
- Greece (9):
  - University General Hospital of Alexandroupolis; Haemotology, Alexandroupoli
  - General Hospital of Athens Evangelismos; Hematology, Athens
  - Laiko General Hospital; Hematology Clinic, Athens
  - Metropolitan Hospital; Hematology Dept, Athens
  - Periph. University General Hospital of Heraklion; Hematology, Heraklion
  - University Hospital of Ioannina; Hematology, Ioannina
  - University Hospital Of Patras; Dept. Of Internal Medicine-Hematology Division, Pátrai
  - Theagenio Anticancer Hospital; Dept. of Haematology, Thessaloniki
  - Georgios Papanikolaou Hospital; Hematology Department, Thessaloniki
- Ireland (5):
  - Cork Uni Hospital; Oncology Dept, Cork
  - Mater Misericordiae Uni Hospital; Oncology, Dublin
  - St James' Hospital; Cancer Clinical Trials Office, Dublin
  - Galway Uni Hospital; Oncology Dept, Galway
  - University Hospital Limerick - Oncology, Limerick
- Israel (9):
  - Haemek Medical Center; Hematology Department, Afula
  - Rambam Medical Center; Heamatology & Bone Marrow Transplantation, Haifa
  - Wolfson Mc; Haematology, Holon
  - Shaare Zedek Medical Center; Hematology Dept., Jerusalem
  - Meir Medical Center; Heamatology Dept, Kfar Saba
  - Beilinson Medical Center; Haematology, Petah Tikva
  - Chaim Sheba Medical Center; Hematology BMT & CBB, Ramat Gan
  - Kaplan Medical Center, Rehovot
  - Ichilov Sourasky Medical Center; Heamatology, Tel Aviv
- Italy (20):
  - Ospedale Civile Dello Spirito Santo; Divisione Di Ematologia, Pescara, Abruzzo
  - Az. Osp. G. Moscati; U.O. Do Ematologia, Taranto, Apulia
  - IRST Istituto Scientifico Romagnolo Per Lo Studio E Cura Dei Tumori, Sede Meldola; Oncologia Medica, Meldola, Emilia-Romagna
  - Az. Osp. S. Maria Delle Croci; U.O. Di Ematologia, Ravenna, Emilia-Romagna
  - Ospedale Infermi Di Rimini; Unità Operativa di Oncologia e Oncoematologia, Rimini, Emilia-Romagna
  - Irccs Centro Di Riferimento Oncologico (CRO); Dipartimento Di Oncologia Medica, Aviano, Friuli Venezia Giulia
  - AOU Ospedali Riuniti; Ematologia, Trieste, Friuli Venezia Giulia
  - Uni Cattolica; Divisione Di Ematologia, Rome, Lazio
  - Az. Osp. Sant'Andrea; U.O. C. Ematologia, Rome, Lazio
  - ASST PAPA GIOVANNI XXIII; Ematologia, Bergamo, Lombardy
  - ASST DI CREMONA; U.O.S. di Ematologia, Cremona, Lombardy
  - Ospedale Di Circolo E Fondazione Macchi; Ematologia, Varese, Lombardy
  - Ospedale Mauriziano Umberto I, Turin, Piedmont
  - Ospedale Oncologico A Businco-Cagliari; Ematologia Sez., Cagliari, Sardinia
  - Azienda Ospedaliero Uni Ria Policlinico G. Martino; U.O. Di Oncologia Medica, Messina, Sicily
  - Casa Di Cura La Maddalena; Oncoematologia E Trapianto Del Midollo Osseo, Palermo, Sicily
  - Ospedale Civile; S.C. Ematologia, Pesaro, The Marches
  - A.O. Univ.Ospedali Riuniti Umerto I -G.M.Lancisi G.Salesi; U.O. Clinica Di Ematologia, Torrette Di Ancona, The Marches
  - Azienda Ospedaliera Di Perugia Ospedale s. Maria Della Misericordia; Oncologia Medica, Perugia, Umbria
  - Uni Degli Studi; Dip.Med.Clinica E Sperim. Ematologia, Padua, Veneto
- Netherlands (16):
  - Medisch Centrum Alkmaar, Alkmaar
  - Meander Medisch Centrum; Locatie Lichtenberg, Amersfoort
  - Deventer Ziekenhuis; Interne Geneeskunde, Deventer
  - Albert Schweitzer Ziekenhuis, Dordrecht
  - Maxima Medisch Centrum; Inwendige Geneeskunde, Eindhoven
  - Groene Hart Ziekenhuis Bleulandlocatie; Inwendige Geneeskunde, Gouda
  - Universitair Medisch Centrum Groningen, Groningen
  - Atrium Medisch Centrum, Heerlen
  - Spaarne Ziekenhuis; Inwendige Geneeskunde, Hoofddorp
  - Medisch Centrum Leeuwarden; Interne, Leeuwarden
  - St. Antonius Ziekenhuis Nieuwegein, Nieuwegein
  - Erasmus Mc - Locatie Centrum; Dept of Hematology, Rotterdam
  - Erasmus Medisch Centrum Rotterdam; Lokatie Daniel den Hoed, Rotterdam
  - Maasstad ziekenhuis, Rotterdam
  - Zuyderland ziekenhuis locatie Geleen, Sittard-Geleen
  - Isala Klinieken, Locatie Sophia; Inwendige Geneeskunde, Zwolle
- Peru (3):
  - Hospital Nacional Almanzor Aguinaga Asenjo; Unidad De Investigacion Del Servicio De Oncologia Medica, Chiclayo
  - Instituto;Oncologico Miraflores, Lima
  - Oncosalud Sac; Oncología, Lima
- Poland (6):
  - Katedra i Klinika Hematologii i Transplantacji Szpiku SUM, Katowice
  - Swietokrzyskie Centrum Onkologii; Onkologia Ogolna, Kielce
  - Malopolskie Centrum Medyczne, Krakow
  - Szpital Wojewodzki w Opolu, Oddzial Hematologii i Onkologii Hematologicznej, Opole
  - Wojewodzki Szpital Specjalistyczny im. J. Korczaka; Oddział Chorób Wewnetrznych/Hematologiczny, Słupsk
  - Centrum Onkologii Instytut im. M. Sklodowskiej-Curie, Klinika Nowotworow Ukladu Chlonnego, Warsaw
- Portugal (5):
  - HUC; Servico de Hematologia, Coimbra
  - Hospital Santo Antonio dos Capuchos; Servico de Hemato-Oncologia, Lisbon
  - Hospital de Santa Maria; Servico de Hematologia e Transplantacao de Medula, Lisbon
  - IPO do Porto; Servico de Onco-Hematologia, Porto
  - Hospital de Sao Joao; Servico de Hematologia Clinica, Porto
- Russia (10):
  - Regional Oncology Center, Chelyabinsk
  - Republican Clinical Oncologic Dispensary of Republic Of Tatarstan, Kazan'
  - N.N.Blokhin Russian Cancer Research Center; Dept. of Chemotherapy & Hemoblastosis, Moscow
  - Rus Med Academy for Postgraduate Education; Oncology Department, Moscow
  - Vladimirskiy Regional Scientific Research Inst. ; Hematology, Moscow
  - Regional Clinical Hospital N.A. Semashko; Hematology, Nizhny Novgorod
  - Clinical MSCh No1, Perm
  - Saint-Petersburg SHI City Clinical Hospital #31, Saint Petersburg
  - City Clinical Hospital #15; Hematology department, Saint Petersburg
  - Central City Hospital #7; Hematology, Yekaterinburg
- Riyadh Military Hospital, Riyadh, Saudi Arabia
- Serbia (2):
  - Clinical Center Kragujevac;Center for Hematology, Kragujevac
  - Clinic of Haematology Cc Nis, Niš
- South Africa (3):
  - National Hospital; Oncotherapy Dept, Bloemfontein
  - Tygerberg Hospital; Haematology Department, Cape Town
  - Steve Biko Academic Hospital; Oncology, Pretoria
- Spain (20):
  - Corporacio Sanitaria Parc Tauli; Servicio de Hematologia, Sabadell, Barcelona
  - Hospital Punta Europa; Servicio de Hematologia, Algeciras, Cadiz
  - Hospital Universitario Marques de Valdecilla; Servicio de Hematologia, Santander, Cantabria
  - Hospital de Donostia; Servicio de Hematologia, Donostia / San Sebastian, Guipuzcoa
  - Hospital de Gran Canaria Dr. Negrin; Servicio de Oncologia, Las Palmas de Gran Canaria, Las Palmas
  - Hospital Universitario Materno Infantil de Gran Canaria; Servicio de Hematologia, Las Palmas de Gran Canarias, Las Palmas
  - Hospital de Cabueñes; Servicio de Hematología y Hemoterapia, Gijón, Principality of Asturias
  - Hospital de Cruces; Servicio de Hematologia, Barakaldo, Vizcaya
  - Hospital General Univ. de Alicante; Servicio de Oncologia, Alicante
  - Hospital Universitari de Girona Dr. Josep Trueta; Servicio de Hematologia, Girona
  - Hospital Lucus Augusti; Servicio de Hematologia, Lugo
  - Hospital General Universitario Gregorio Marañon; Servicio de Hematología, Madrid
  - Hospital Univ. 12 de Octubre; Servicio de Hematologia, Madrid
  - Hospital Universitario la Paz; Servicio de Hematologia, Madrid
  - Hospital Universitario Puerta de Hierro; Servicio de Oncologia, Madrid
  - Hospital Costa del Sol; Servicio de Hematologia, Málaga
  - Hospital Clinico Universitario de Valencia; Servicio de Onco-hematologia, Valencia
  - Hospital Universitario Dr. Peset; Servicio de Hematologia, Valencia
  - Hospital Clinico Universitario Lozano Blesa; Servicio de Hematologia, Zaragoza
  - Hospital Universitario Miguel Servet; Servicio Hematologia, Zaragoza
- Thailand (4):
  - King Chulalongkorn Memorial Hospital; Division of Hematology, Department of Medicine, Bangkok
  - Ramathibodi Hospital; Division of Hematology, Department of Medicine, Bangkok
  - Siriraj Hospital; Division of Hematology, Department of Medicine, Bangkok
  - Srinagarind Hospital, Khon Kaen Uni ; Dept of Medicine, Khon Kaen
- Turkey (Türkiye) (12):
  - Cukurova Uni ; Hematology, Adana
  - Diskapi Research And Training Hospital; hematology, Ankara
  - Hacettepe Uni Medical Faculty; Hematology, Ankara
  - Ankara University; Hematology, Ankara
  - Gaziantep Uni Medical School; Hematology, Gaziantep
  - Istanbul University Cerrahpasa Medical Faculty; Hematology Department, Istanbul
  - Dokuz Eylul Uni ; Hematology, Izmir
  - Ege Uni Medical School; Hematology, Izmir
  - Erciyes Uni ; Hematology, Kayseri
  - Ondokuzmayis University Medical Faculty Heamatology Department, Samsun
  - Cumhuriyet Uni. Med. Fac.; Hematology, Sivas
  - Karadeniz Technical Uni School of Medicine; Hematology, Trabzon
- Ukraine (3):
  - Mun. Multifield Clin.Hosp.#4,Dept. of Chemotherapy, DSMU; Chair of Oncology and Medical Radiology, Dnipropetrovsk
  - Kyiv City Clinical Oncological Center; Chemotherapy Department, Kiev
  - State Oncology Regional Treatment-Diagnostic Center; Chemotherapy Department, Lviv
- United Kingdom (5):
  - SOUTHMEAD HOSPITAL; Richard Bright Dialysis Centre, Bristol
  - Ipswich Hospital; Oncology Pharmacy, Ipswich
  - Macclesfield District General Hospital, Macclesfield
  - Kings Mill Hospital, Sutton in Ashfield
  - Singleton Hospital: Pharmacy Department, Swansea
- Venezuela (2):
  - Instituto de Oncologia y Hematologia UCV, Caracas
  - Banco Municipal de Sangre; Hematología, Caracas

REFERENCES:
- [Derived] Lugtenburg P, Avivi I, Berenschot H, Ilhan O, Marolleau JP, Nagler A, Rueda A, Tani M, Turgut M, Osborne S, Smith R, Pfreundschuh M. Efficacy and safety of subcutaneous and intravenous rituximab plus cyclophosphamide, doxorubicin, vincristine, and prednisone in first-line diffuse large B-cell lymphoma: the randomized MabEase study. Haematologica. 2017 Nov;102(11):1913-1922. doi: 10.3324/haematol.2017.173583. Epub 2017 Sep 21. PMID 28935843

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 662 individuals were screened for entry into the study, and 86 failed the screening procedure. Overall, 576 participants were randomized; 572 received treatment and were included in the analyses.
Groups:
- Rituximab Subcutaneous (SC): Participants with previously untreated, cluster of differentiation (CD) 20-positive diffuse large B-cell lymphoma (DLBCL) received up to 8 cycles of rituximab in combination with cyclophosphamide, doxorubicin, vincristine, and prednisone (CHOP). Treatment was given on Day 1 of each cycle, and the cycle length (14 or 21 days) was decided by the study center. For Cycle 1, rituximab was administered at a dose of 375 milligrams per meter-squared (mg/m^2) via IV infusion; subsequent doses were given as 1400 milligrams (mg) via SC injection. Tumor response was assessed after 4 cycles according to criteria published by Cheson et al (1999), which are presented in Outcome Measure 1. The duration of CHOP therapy could be reduced from 8 to 6 cycles for those who achieved complete response (CR) or complete response unconfirmed (CRu) after 4 cycles, but all participants received a full 8 cycles of rituximab.
- Rituximab Intravenous (IV): Participants with previously untreated, CD20-positive DLBCL received up to 8 cycles of rituximab in combination with CHOP. Treatment was given on Day 1 of each cycle, and the cycle length (14 or 21 days) was decided by the study center. For all cycles, rituximab was administered at a dose of 375 mg/m^2 via IV infusion. Tumor response was assessed after 4 cycles according to criteria published by Cheson et al (1999), which are presented in Outcome Measure 1. The duration of CHOP therapy could be reduced from 8 to 6 cycles for those who achieved CR or CRu after 4 cycles, but all participants received a full 8 cycles of rituximab.
Period: Overall Study
Arm/Group | Rituximab Subcutaneous (SC) | Rituximab Intravenous (IV)
Started | 369 | 203
Completed | 230 | 125
Not Completed | 139 | 78
Not completed — Withdrawal by Subject | 14 | 14
Not completed — Protocol Violation | 4 | 4
Not completed — Treatment Failure | 1 | 1
Not completed — Death | 69 | 34
Not completed — Stable or Progressed Disease | 5 | 3
Not completed — Lost to Follow-up | 20 | 16
Not completed — Lack of Compliance | 6 | 1
Not completed — Other | 20 | 5

BASELINE CHARACTERISTICS:
Population: Safety Population: All participants who received at least one dose of study drug according to treatment received.
Groups:
- Rituximab SC: Participants with previously untreated, CD20-positive DLBCL received up to 8 cycles of rituximab in combination with CHOP. Treatment was given on Day 1 of each cycle, and the cycle length (14 or 21 days) was decided by the study center. For Cycle 1, rituximab was administered at a dose of 375 mg/m^2 via IV infusion; subsequent doses were given as 1400 mg via SC injection. Tumor response was assessed after 4 cycles according to criteria published by Cheson et al (1999), which are presented in Outcome Measure 1. The duration of CHOP therapy could be reduced from 8 to 6 cycles for those who achieved CR or CRu after 4 cycles, but all participants received a full 8 cycles of rituximab.
- Rituximab IV: Participants with previously untreated, CD20-positive DLBCL received up to 8 cycles of rituximab in combination with CHOP. Treatment was given on Day 1 of each cycle, and the cycle length (14 or 21 days) was decided by the study center. For all cycles, rituximab was administered at a dose of 375 mg/m^2 via IV infusion. Tumor response was assessed after 4 cycles according to criteria published by Cheson et al (1999), which are presented in Outcome Measure 1. The duration of CHOP therapy could be reduced from 8 to 6 cycles for those who achieved CR or CRu after 4 cycles, but all participants received a full 8 cycles of rituximab.
- Total: Total of all reporting groups
Arm/Group | Rituximab SC | Rituximab IV | Total
Number analyzed (Participants) | 369 | 203 | 572
Age, Continuous [Mean (Standard Deviation); unit: years] | 60.4 (13.78) | 61.0 (12.63) | 60.6 (13.38)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 165 | 100 | 265
  Male | 204 | 103 | 307

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Complete Response (CR) or Complete Response Unconfirmed (CRu)
Description: Tumor response was assessed per criteria published by Cheson et al (1999). According to consensus recommendations, CR was defined as complete disappearance of all clinical and radiographic evidence of disease and disease-related symptoms, regression of lymph nodes to normal size, absence of splenomegaly, and absence of bone marrow involvement. CRu was defined as disappearance of clinical and radiographic evidence of disease and absence of splenomegaly, with regression of lymph nodes by greater than (>) 75 percent (%) but still >1.5 centimeters (cm) in size, and indeterminate bone marrow assessment. The percentage of participants with either response at the end of induction (EOI) was determined with corresponding 95% Pearson-Clopper confidence interval (CI).
Time Frame: Up to approximately 4.25 years
Population: Intent-to-Treat (ITT) Population: All participants who completed Baseline and at least one on-treatment efficacy assessment.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Rituximab SC | Rituximab IV
Number analyzed (Participants) | 342 | 177
percentage of participants | 50.6 [45.2 to 56.0] | 42.4 [35.0 to 50.0]
Statistical Analysis 1: Comparison: Rituximab SC vs Rituximab IV; Test type: Superiority or Other; p = 0.076, Chi-squared; Difference in Response Rates = 8.2, 95% CI [-1.1 to 17.5]

2. Secondary Outcome: Cancer Treatment Satisfaction Questionnaire (CTSQ) Domain Scores
Description: The CTSQ is a validated 16-item questionnaire that measures three domains related to satisfaction with cancer therapy. These include expectations of therapy, feelings about side effects, and satisfaction with therapy. Each domain is scored on a scale of 0 to 100, with higher scores indicative of more positive feelings toward therapy. The score for each domain was averaged among all participants.
Time Frame: At Cycle 7 (each cycle was 14 or 21 days)
Population: ITT Population (CTSQ Subpopulation): All participants who completed the CTSQ at Cycles 3 and 7; number (n) = number of participants in the analysis for the specified domain.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Rituximab SC | Rituximab IV
Number analyzed (Participants) | 280 | 141
units on a scale
  Expectations of Therapy (n=280,141) | 79.35 (17.422) | 82.94 (16.536)
  Feelings about Side Effects (n=276,141) | 60.69 (21.594) | 57.62 (23.339)
  Satisfaction with Therapy (n=278,141) | 85.92 (11.428) | 83.60 (13.451)

3. Secondary Outcome: Rituximab Administration Satisfaction Questionnaire (RASQ) Domain Scores
Description: The RASQ is a 20-item questionnaire that measures five domains related to the impact of treatment administration. These include physical impact, psychological impact, impact on activities of daily living (ADLs), convenience, and satisfaction. Each domain is scored on a scale of 0 to 100, with higher scores indicative of more positive feelings toward therapy. The score for each domain was averaged among all participants.
Time Frame: At Cycle 7 (each cycle was 14 or 21 days)
Population: ITT Population (RASQ Subpopulation): All participants who completed the RASQ at Cycles 3 and 7; n = number of participants in the analysis for the specified domain.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Rituximab SC | Rituximab IV
Number analyzed (Participants) | 284 | 144
units on a scale
  Physical Impact (n=278,140) | 86.24 (14.012) | 81.49 (16.848)
  Psychological Impact (n=277,141) | 85.65 (13.920) | 78.65 (18.233)
  Impact on ADLs (n=266,140) | 83.77 (16.117) | 57.38 (19.230)
  Convenience (n=279,143) | 82.32 (13.428) | 60.14 (17.473)
  Satisfaction (n=282,141) | 89.58 (12.051) | 77.39 (18.232)

4. Secondary Outcome: Median Duration of Rituximab Administration for Each Treatment Cycle
Description: Duration of rituximab administration was defined as the time from start to end of the SC injection or IV infusion. The median duration was reported.
Time Frame: Cycles 1, 2, 3, 4, 5, 6, 7, and 8 (each cycle was 14 or 21 days)
Population: Safety Population; n = number of participants in the analysis for the specified timepoint.
Measure: Median (Full Range); unit: hours
Arm/Group | Rituximab SC | Rituximab IV
Number analyzed (Participants) | 369 | 203
hours
  Cycle 1 (n=346,190) | 4.0 [0.10 to 11.00] | 4.0 [1.20 to 10.00]
  Cycle 2 (n=361,178) | 0.1 [0.10 to 23.10] | 3.0 [0.50 to 10.00]
  Cycle 3 (n=349,177) | 0.1 [0.10 to 5.50] | 2.8 [1.00 to 21.40]
  Cycle 4 (n=346,173) | 0.1 [0.00 to 2.50] | 2.7 [0.50 to 8.00]
  Cycle 5 (n=332,165) | 0.1 [0.00 to 2.50] | 2.6 [0.10 to 8.10]
  Cycle 6 (n=319,162) | 0.1 [0.00 to 2.50] | 2.7 [0.10 to 20.00]
  Cycle 7 (n=304,156) | 0.1 [0.00 to 23.60] | 2.7 [0.50 to 6.70]
  Cycle 8 (n=305,152) | 0.1 [0.00 to 2.50] | 2.55 [0.10 to 17.90]
  Overall (n=368,201) | 4.7 [0.10 to 28.70] | 19.00 [1.20 to 57.40]

5. Secondary Outcome: Percentage of Participants by Time Spent in the Infusion Chair/Bed for Each Treatment Cycle
Description: Chair time was defined as the amount of time the participant occupied an infusion chair/bed for a single treatment cycle of rituximab + CHOP chemotherapy. Where the chair time was not documented for a given cycle, it was reported as "Missing".
Time Frame: Cycles 1, 2, 3, 4, 5, 6, 7, and 8 (each cycle was 14 or 21 days)
Population: Safety Population.
Measure: Number; unit: percentage of participants
Arm/Group | Rituximab SC | Rituximab IV
Number analyzed (Participants) | 369 | 203
percentage of participants
  Less than 30 minutes (Cycle 1) | 0 | 0
  30 minutes to 1 hour (Cycle 1) | 0 | 0.5
  1 to 2 hours (Cycle 1) | 1.4 | 0
  2 to 4 hours (Cycle 1) | 20.6 | 17.2
  4 to 12 hours (Cycle 1) | 69.4 | 72.4
  More than 12 hours (Cycle 1) | 7.3 | 7.9
  Missing (Cycle 1) | 1.4 | 2.0
  Less than 30 minutes (Cycle 2) | 7.3 | 0
  30 minutes to 1 hour (Cycle 2) | 2.4 | 0
  1 to 2 hours (Cycle 2) | 17.1 | 1.1
  2 to 4 hours (Cycle 2) | 56.1 | 36.2
  4 to 12 hours (Cycle 2) | 12.2 | 60.1
  More than 12 hours (Cycle 2) | 0.3 | 1.1
  Missing (Cycle 2) | 4.6 | 1.6
  Less than 30 minutes (Cycle 3) | 5.6 | 0
  30 minutes to 1 hour (Cycle 3) | 2.0 | 0
  1 to 2 hours (Cycle 3) | 22.1 | 0.5
  2 to 4 hours (Cycle 3) | 55.9 | 38.9
  4 to 12 hours (Cycle 3) | 12.6 | 58.4
  More than 12 hours (Cycle 3) | 0.3 | 0.5
  Missing (Cycle 3) | 1.7 | 1.6
  Less than 30 minutes (Cycle 4) | 5.1 | 0
  30 minutes to 1 hour (Cycle 4) | 2.8 | 0
  1 to 2 hours (Cycle 4) | 21.8 | 1.1
  2 to 4 hours (Cycle 4) | 55.0 | 36.7
  4 to 12 hours (Cycle 4) | 13.9 | 60.6
  More than 12 hours (Cycle 4) | 0.3 | 0.6
  Missing (Cycle 4) | 1.1 | 1.1
  Less than 30 minutes (Cycle 5) | 5.0 | 0.6
  30 minutes to 1 hour (Cycle 5) | 2.4 | 0
  1 to 2 hours (Cycle 5) | 25.2 | 1.1
  2 to 4 hours (Cycle 5) | 53.4 | 40.2
  4 to 12 hours (Cycle 5) | 12.8 | 56.3
  More than 12 hours (Cycle 5) | 0 | 0.6
  Missing (Cycle 5) | 1.2 | 1.1
  Less than 30 minutes (Cycle 6) | 3.4 | 0.6
  30 minutes to 1 hour (Cycle 6) | 3.1 | 0
  1 to 2 hours (Cycle 6) | 23.0 | 1.8
  2 to 4 hours (Cycle 6) | 56.7 | 42.5
  4 to 12 hours (Cycle 6) | 12.3 | 53.3
  More than 12 hours (Cycle 6) | 0 | 0
  Missing (Cycle 6) | 1.5 | 1.8
  Less than 30 minutes (Cycle 7) | 18.7 | 0
  30 minutes to 1 hour (Cycle 7) | 7.0 | 0
  1 to 2 hours (Cycle 7) | 26.9 | 4.9
  2 to 4 hours (Cycle 7) | 40.2 | 48.8
  4 to 12 hours (Cycle 7) | 6.0 | 44.4
  More than 12 hours (Cycle 7) | 0 | 0
  Missing (Cycle 7) | 1.3 | 1.9
  Less than 30 minutes (Cycle 8) | 20.3 | 0.6
  30 minutes to 1 hour (Cycle 8) | 6.4 | 0
  1 to 2 hours (Cycle 8) | 29.3 | 4.4
  2 to 4 hours (Cycle 8) | 36.7 | 50.9
  4 to 12 hours (Cycle 8) | 5.8 | 43.4
  More than 12 hours (Cycle 8) | 0 | 0
  Missing (Cycle 8) | 1.6 | 0.6

6. Secondary Outcome: Percentage of Participants by Time Spent in the Hospital for Each Treatment Cycle
Description: Hospital time was defined as the amount of time the participant was in the hospital for the course of one cycle of rituximab + CHOP chemotherapy. Where the hospital time was not documented for a given cycle, it was reported as "Missing".
Time Frame: Cycles 1, 2, 3, 4, 5, 6, 7, and 8 (each cycle was 14 or 21 days)
Population: Safety Population.
Measure: Number; unit: percentage of participants
Arm/Group | Rituximab SC | Rituximab IV
Number analyzed (Participants) | 369 | 203
percentage of participants
  Less than 2 hours (Cycle 1) | 0.3 | 0
  2 to 4 hours (Cycle 1) | 3.0 | 1.5
  4 to 6 hours (Cycle 1) | 19.8 | 20.7
  6 to 12 hours (Cycle 1) | 39.0 | 43.8
  12 to 24 hours (Cycle 1) | 8.9 | 6.9
  More than 24 hours (Cycle 1) | 26.8 | 24.1
  Missing (Cycle 1) | 2.2 | 3.0
  Less than 2 hours (Cycle 2) | 3.8 | 0
  2 to 4 hours (Cycle 2) | 33.1 | 10.1
  4 to 6 hours (Cycle 2) | 27.9 | 33.5
  6 to 12 hours (Cycle 2) | 16.3 | 38.8
  12 to 24 hours (Cycle 2) | 3.8 | 1.1
  More than 24 hours (Cycle 2) | 10.3 | 11.7
  Missing (Cycle 2) | 4.9 | 4.8
  Less Than 2 hours (Cycle 3) | 3.6 | 0.5
  2 to 4 hours (Cycle 3) | 37.2 | 11.9
  4 to 6 hours (Cycle 3) | 30.2 | 30.8
  6 to 12 hours (Cycle 3) | 14.5 | 41.6
  12 to 24 hours (Cycle 3) | 2.8 | 2.2
  More than 24 hours (Cycle 3) | 9.8 | 10.3
  Missing (Cycle 3) | 2.0 | 2.7
  Less Than 2 hours (Cycle 4) | 4.5 | 0
  2 to 4 hours (Cycle 4) | 36.3 | 10.0
  4 to 6 hours (Cycle 4) | 27.5 | 31.1
  6 to 12 hours (Cycle 4) | 17.6 | 42.2
  12 to 24 hours (Cycle 4) | 2.0 | 2.8
  More than 24 hours (Cycle 4) | 10.2 | 10.6
  Missing (Cycle 4) | 2.0 | 3.3
  Less Than 2 hours (Cycle 5) | 5.0 | 0.6
  2 to 4 hours (Cycle 5) | 39.5 | 11.5
  4 to 6 hours (Cycle 5) | 26.4 | 34.5
  6 to 12 hours (Cycle 5) | 16.0 | 37.4
  12 to 24 hours (Cycle 5) | 2.1 | 1.7
  More than 24 hours (Cycle 5) | 8.9 | 10.9
  Missing (Cycle 5) | 2.1 | 3.4
  Less Than 2 hours (Cycle 6) | 4.3 | 0.6
  2 to 4 hours (Cycle 6) | 39.6 | 12.6
  4 to 6 hours (Cycle 6) | 26.4 | 34.1
  6 to 12 hours (Cycle 6) | 16.3 | 38.3
  12 to 24 hours (Cycle 6) | 2.5 | 2.4
  More than 24 hours (Cycle 6) | 8.6 | 9.0
  Missing (Cycle 6) | 2.5 | 3.0
  Less Than 2 hours (Cycle 7) | 17.7 | 0
  2 to 4 hours (Cycle 7) | 40.8 | 23.5
  4 to 6 hours (Cycle 7) | 19.9 | 36.4
  6 to 12 hours (Cycle 7) | 10.4 | 30.9
  12 to 24 hours (Cycle 7) | 2.8 | 2.5
  More than 24 hours (Cycle 7) | 5.7 | 3.7
  Missing (Cycle 7) | 2.5 | 3.1
  Less Than 2 hours (Cycle 8) | 18.0 | 0
  2 to 4 hours (Cycle 8) | 40.5 | 25.8
  4 to 6 hours (Cycle 8) | 21.9 | 34.0
  6 to 12 hours (Cycle 8) | 8.7 | 30.8
  12 to 24 hours (Cycle 8) | 2.6 | 1.3
  More than 24 hours (Cycle 8) | 5.8 | 5.0
  Missing (Cycle 8) | 2.6 | 3.1

7. Secondary Outcome: Number of Participants With an Event-Free Survival (EFS) Event
Description: EFS events included disease progression, relapse, initiation of other anti-lymphoma therapy, or death. Tumor response was assessed according to criteria published by Cheson et al (1999). Progression was defined as greater than or equal to (≥) 50% increase in the sum of products of greatest diameters of any previously identified abnormal lymph node or the appearance of any new lesion. Relapse was defined as a new lesion or increase by ≥50% in size of previously involved sites, or ≥50% increase in greatest diameter of any previously identified node >1 cm, following an earlier assessment of CR or CRu.
Time Frame: Up to approximately 4.25 years
Population: ITT Population.
Measure: Number; unit: participants
Arm/Group | Rituximab SC | Rituximab IV
Number analyzed (Participants) | 342 | 177
participants | 116 | 53

8. Secondary Outcome: Duration of EFS
Description: EFS was defined as the time from randomization to first occurrence of disease progression, relapse, initiation of other anti-lymphoma therapy, or death, whichever occurred first. Tumor response was assessed according to criteria published by Cheson et al (1999). Progression was defined as a ≥50% increase in the sum of products of greatest diameters of any previously identified abnormal lymph node or the appearance of any new lesion. Relapse was defined as a new lesion or increase by ≥50% in size of previously involved sites, or ≥50% increase in greatest diameter of any previously identified node >1 cm, following an earlier assessment of CR or CRu.
Time Frame: Up to approximately 4.25 years
Population: ITT Population.
Measure: Median (Full Range); unit: months
Arm/Group | Rituximab SC | Rituximab IV
Number analyzed (Participants) | 342 | 177
months | NA [NA to NA] — Median EFS was not reached. | NA [NA to NA] — Median EFS was not reached.

9. Secondary Outcome: Number of Participants With Relapse or Death at the Time of Primary Analysis
Description: Tumor response was assessed according to criteria published by Cheson et al (1999). Relapse was defined as a new lesion or increase by ≥50% in size of previously involved sites, or ≥50% increase in greatest diameter of any previously identified node >1 cm, following an earlier assessment of CR or CRu. The number of participants who had experienced relapse or death prior to the clinical cut-off date (October 2014) was determined.
Time Frame: Up to approximately 2 years (assessed at Baseline, Day 1 of each cycle [maximum 8 cycles; each cycle was 14 or 21 days], every 3 months thereafter, and/or 4 weeks after early termination)
Population: ITT Population (Responder Subpopulation): All participants who achieved CR or CRu after 4 cycles.
Measure: Number; unit: participants
Arm/Group | Rituximab SC | Rituximab IV
Number analyzed (Participants) | 178 | 90
participants | 12 | 5

10. Secondary Outcome: Duration of Disease-Free Survival (DFS)
Description: DFS was defined as the time from date of initial CR/CRu to the date of relapse or death from any cause. Tumor response was assessed according to criteria published by Cheson et al (1999). Relapse was defined as a new lesion or increase by ≥50% in size of previously involved sites, or ≥50% increase in greatest diameter of any previously identified node >1 cm, following an earlier assessment of CR or CRu.
Time Frame: Up to approximately 4.25 years
Population: ITT Population (Responder Subpopulation).
Measure: Median (Full Range); unit: months
Arm/Group | Rituximab SC | Rituximab IV
Number analyzed (Participants) | 240 | 118
months | NA [NA to NA] — Median DFS was not reached. | NA [NA to NA] — Median DFS was not reached.

11. Secondary Outcome: Number of Participants With Progression, Relapse, or Death
Description: Tumor response was assessed according to criteria published by Cheson et al (1999). Progression was defined as ≥50% increase in the sum of products of greatest diameters of any previously identified abnormal lymph node or the appearance of any new lesion. Relapse was defined as a new lesion or increase by ≥50% in size of previously involved sites, or ≥50% increase in greatest diameter of any previously identified node >1 cm, following an earlier assessment of CR or CRu.
Time Frame: Up to approximately 4.25 years
Population: ITT Population.
Measure: Number; unit: participants
Arm/Group | Rituximab SC | Rituximab IV
Number analyzed (Participants) | 342 | 177
participants | 95 | 38

12. Secondary Outcome: Duration of Progression-Free Survival (PFS)
Description: PFS was defined as the time from randomization to first occurrence of disease progression, relapse, or death from any cause. Tumor response was assessed according to criteria published by Cheson et al (1999). Progression was defined as ≥50% increase in the sum of products of greatest diameters of any previously identified abnormal lymph node or the appearance of any new lesion. Relapse was defined as a new lesion or increase by ≥50% in size of previously involved sites, or ≥50% increase in greatest diameter of any previously identified node >1 cm, following an earlier assessment of CR or CRu.
Time Frame: Up to approximately 4.25 years
Population: ITT Population.
Measure: Median (Full Range); unit: months
Arm/Group | Rituximab SC | Rituximab IV
Number analyzed (Participants) | 342 | 177
months | NA [NA to NA] — Median PFS was not reached. | NA [NA to NA] — Median PFS was not reached.

13. Secondary Outcome: Number of Deaths
Time Frame: Up to approximately 4.25 years
Population: ITT Population.
Measure: Number; unit: participants
Arm/Group | Rituximab SC | Rituximab IV
Number analyzed (Participants) | 342 | 177
participants | 56 | 22

14. Secondary Outcome: Duration of Overall Survival (OS)
Description: OS was defined as the time from randomization to death from any cause.
Time Frame: Up to approximately 4.25 years
Population: ITT Population.
Measure: Median (Full Range); unit: months
Arm/Group | Rituximab SC | Rituximab IV
Number analyzed (Participants) | 342 | 177
months | NA [NA to NA] — Median OS was not reached. | NA [NA to NA] — Median OS was not reached.

ADVERSE EVENTS:
Time Frame: Up to approximately 4.25 years
Description: Safety Population.
Arm/Group | Rituximab SC | Rituximab IV
Serious Adverse Events (participants affected / at risk) | 155/369 | 77/203
Other Adverse Events (participants affected / at risk) | 319/369 | 172/203
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Rituximab SC (N=369) | Rituximab IV (N=203)
Febrile neutropenia (Blood and lymphatic system disorders) | 49 | 24
Neutropenia (Blood and lymphatic system disorders) | 22 | 10
Anaemia (Blood and lymphatic system disorders) | 2 | 2
Leukopenia (Blood and lymphatic system disorders) | 1 | 3
Febrile bone marrow aplasia (Blood and lymphatic system disorders) | 0 | 1
Pancytopenia (Blood and lymphatic system disorders) | 1 | 0
Pneumonia (Infections and infestations) | 27 | 7
Septic shock (Infections and infestations) | 3 | 3
Lung infection (Infections and infestations) | 4 | 1
Respiratory tract infection (Infections and infestations) | 2 | 0
Sepsis (Infections and infestations) | 5 | 0
Cellulitis (Infections and infestations) | 2 | 0
Infection (Infections and infestations) | 2 | 0
Lower respiratory tract infection (Infections and infestations) | 1 | 1
Urosepsis (Infections and infestations) | 1 | 1
Anal abscess (Infections and infestations) | 1 | 0
Appendicitis (Infections and infestations) | 2 | 0
Bronchiolitis (Infections and infestations) | 1 | 0
Bronchitis (Infections and infestations) | 1 | 0
Clostridium difficile colitis (Infections and infestations) | 1 | 0
Erysipelas (Infections and infestations) | 1 | 0
Gastroenteritis (Infections and infestations) | 1 | 0
H1N1 influenza (Infections and infestations) | 1 | 0
Herpes oesophagitis (Infections and infestations) | 1 | 0
Herpes simplex hepatitis (Infections and infestations) | 1 | 0
Herpes zoster (Infections and infestations) | 2 | 0
Klebsiella sepsis (Infections and infestations) | 1 | 0
Neutropenic infection (Infections and infestations) | 1 | 0
Oral candidiasis (Infections and infestations) | 1 | 0
Oral herpes (Infections and infestations) | 1 | 0
Peritonitis (Infections and infestations) | 1 | 0
Pneumocystis jirovecii infection (Infections and infestations) | 0 | 1
Pneumocystis jirovecii pneumonia (Infections and infestations) | 1 | 0
Sinusitis (Infections and infestations) | 0 | 1
Tuberculosis (Infections and infestations) | 0 | 1
Upper respiratory tract infection (Infections and infestations) | 1 | 0
Urinary tract infection (Infections and infestations) | 1 | 1
Viral infection (Infections and infestations) | 0 | 1
Viral upper respiratory tract infection (Infections and infestations) | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 3 | 1
Diarrhoea (Gastrointestinal disorders) | 2 | 0
Vomiting (Gastrointestinal disorders) | 3 | 0
Nausea (Gastrointestinal disorders) | 1 | 1
Abdominal distension (Gastrointestinal disorders) | 1 | 0
Anal fissure (Gastrointestinal disorders) | 1 | 0
Anal haemorrhage (Gastrointestinal disorders) | 1 | 0
Constipation (Gastrointestinal disorders) | 0 | 1
Gastric perforation (Gastrointestinal disorders) | 0 | 1
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 0
Haematemesis (Gastrointestinal disorders) | 1 | 0
Haemorrhoidal haemorrhage (Gastrointestinal disorders) | 1 | 0
Ileus (Gastrointestinal disorders) | 2 | 0
Intestinal obstruction (Gastrointestinal disorders) | 1 | 0
Large intestine perforation (Gastrointestinal disorders) | 1 | 0
Neutropenic colitis (Gastrointestinal disorders) | 1 | 0
Obstruction gastric (Gastrointestinal disorders) | 1 | 0
Pancreatitis (Gastrointestinal disorders) | 1 | 0
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 2 | 0
Pyrexia (General disorders) | 7 | 3
Chills (General disorders) | 2 | 2
Chest pain (General disorders) | 0 | 1
Death (General disorders) | 2 | 0
Fatigue (General disorders) | 0 | 1
General physical health deterioration (General disorders) | 1 | 0
Influenza like illness (General disorders) | 0 | 1
Injection site hypertrophy (General disorders) | 1 | 0
Localised oedema (General disorders) | 0 | 1
Mucosal inflammation (General disorders) | 1 | 0
Oedema peripheral (General disorders) | 1 | 0
Sudden death (General disorders) | 0 | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 | 3
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 1 | 2
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 3
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 2 | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Organising pneumonia (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pleurisy (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pulmonary fibrosis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Atrial fibrillation (Cardiac disorders) | 2 | 3
Cardiac arrest (Cardiac disorders) | 1 | 3
Atrial flutter (Cardiac disorders) | 1 | 1
Myocardial infarction (Cardiac disorders) | 0 | 2
Tachycardia (Cardiac disorders) | 1 | 1
Acute myocardial infarction (Cardiac disorders) | 1 | 0
Cardiac failure (Cardiac disorders) | 1 | 0
Cardiac failure acute (Cardiac disorders) | 1 | 0
Congestive cardiomyopathy (Cardiac disorders) | 1 | 0
Left ventricular failure (Cardiac disorders) | 1 | 0
Sinus tachycardia (Cardiac disorders) | 0 | 1
Supraventricular tachycardia (Cardiac disorders) | 1 | 0
Tachycardia induced cardiomyopathy (Cardiac disorders) | 1 | 0
Neutrophil count decreased (Investigations) | 3 | 3
White blood cell count decreased (Investigations) | 1 | 0
Hepatic enzyme increased (Investigations) | 1 | 0
Troponin T increased (Investigations) | 1 | 0
Weight decreased (Investigations) | 1 | 0
Syncope (Nervous system disorders) | 2 | 1
Cerebrovascular accident (Nervous system disorders) | 2 | 1
Presyncope (Nervous system disorders) | 2 | 0
Cerebral infarction (Nervous system disorders) | 0 | 1
Dysarthria (Nervous system disorders) | 0 | 1
Multiple fractures (Injury, poisoning and procedural complications) | 2 | 0
Femur fracture (Injury, poisoning and procedural complications) | 2 | 0
Fracture (Injury, poisoning and procedural complications) | 0 | 1
Hip fracture (Injury, poisoning and procedural complications) | 0 | 1
Infusion related reaction (Injury, poisoning and procedural complications) | 0 | 1
Lower limb fracture (Injury, poisoning and procedural complications) | 1 | 0
Subdural haematoma (Injury, poisoning and procedural complications) | 0 | 1
Transfusion reaction (Injury, poisoning and procedural complications) | 0 | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 1 | 1
Hyponatraemia (Metabolism and nutrition disorders) | 2 | 0
Dehydration (Metabolism and nutrition disorders) | 1 | 0
Diabetes mellitus inadequate control (Metabolism and nutrition disorders) | 0 | 1
Deep vein thrombosis (Vascular disorders) | 1 | 0
Embolism venous (Vascular disorders) | 1 | 0
Flushing (Vascular disorders) | 0 | 1
Hypotension (Vascular disorders) | 0 | 1
Orthostatic hypotension (Vascular disorders) | 0 | 1
Subclavian vein thrombosis (Vascular disorders) | 0 | 1
Thrombosis (Vascular disorders) | 0 | 1
Bone pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 0
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 0 | 1
Pathological fracture (Musculoskeletal and connective tissue disorders) | 0 | 1
Tendonitis (Musculoskeletal and connective tissue disorders) | 1 | 0
Papillary thyroid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Renal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Transitional cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Adjustment disorder (Psychiatric disorders) | 1 | 0
Anxiety (Psychiatric disorders) | 1 | 0
Confusional state (Psychiatric disorders) | 0 | 1
Depression (Psychiatric disorders) | 1 | 0
Bile duct obstruction (Hepatobiliary disorders) | 1 | 0
Proteinuria (Renal and urinary disorders) | 1 | 0
Prostatitis (Reproductive system and breast disorders) | 1 | 0
Hypernatraemia (Metabolism and nutrition disorders) | 0 | 1
Gastroenteritis norovirus (Infections and infestations) | 1 | 0
Intervertebral discitis (Infections and infestations) | 1 | 0
Localised infection (Infections and infestations) | 1 | 0
Lower respiratory tract infection viral (Infections and infestations) | 1 | 1
Pneumonia cytomegaloviral (Infections and infestations) | 1 | 0
Inguinal hernia (Gastrointestinal disorders) | 0 | 1
Small intestinal perforation (Gastrointestinal disorders) | 1 | 0
Ill-defined disorder (General disorders) | 1 | 0
Cardiac failure congestive (Cardiac disorders) | 1 | 1
Acute coronary syndrome (Cardiac disorders) | 0 | 1
Ischaemic stroke (Nervous system disorders) | 1 | 0
Seizure (Nervous system disorders) | 0 | 1
Transient ischaemic attack (Nervous system disorders) | 0 | 1
Alanine aminotransferase increased (Investigations) | 1 | 0
Blood bilirubin increased (Investigations) | 1 | 0
Platelet count decreased (Investigations) | 1 | 0
Procedural pneumothorax (Injury, poisoning and procedural complications) | 1 | 0
Non-small cell lung cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0
Invasive ductal breast carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Lung adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Metastatic renal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Myelodysplastic syndrome (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Prostate cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Arterial disorder (Vascular disorders) | 1 | 0
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 | 0
Spondylolisthesis (Musculoskeletal and connective tissue disorders) | 1 | 0
Cholecystitis (Hepatobiliary disorders) | 0 | 1
Hepatic failure (Hepatobiliary disorders) | 1 | 0
Haematuria (Renal and urinary disorders) | 1 | 0
Urinary retention (Renal and urinary disorders) | 0 | 1
Cytokine release syndrome (Immune system disorders) | 0 | 1
Eczema (Skin and subcutaneous tissue disorders) | 1 | 0
Knee arthroplasty (Surgical and medical procedures) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Rituximab SC (N=369) | Rituximab IV (N=203)
Neutropenia (Blood and lymphatic system disorders) | 104 | 54
Anaemia (Blood and lymphatic system disorders) | 88 | 40
Nausea (Gastrointestinal disorders) | 79 | 47
Constipation (Gastrointestinal disorders) | 56 | 34
Diarrhoea (Gastrointestinal disorders) | 52 | 20
Vomiting (Gastrointestinal disorders) | 40 | 17
Stomatitis (Gastrointestinal disorders) | 23 | 11
Abdominal pain (Gastrointestinal disorders) | 24 | 12
Fatigue (General disorders) | 71 | 29
Pyrexia (General disorders) | 40 | 23
Asthenia (General disorders) | 42 | 24
Mucosal inflammation (General disorders) | 29 | 16
Oedema peripheral (General disorders) | 27 | 9
Alopecia (Skin and subcutaneous tissue disorders) | 87 | 48
Neuropathy peripheral (Nervous system disorders) | 44 | 24
Paraesthesia (Nervous system disorders) | 32 | 13
Headache (Nervous system disorders) | 21 | 15
Neutrophil count decreased (Investigations) | 81 | 43
Weight decreased (Investigations) | 28 | 8
White blood cell count decreased (Investigations) | 51 | 23
Cough (Respiratory, thoracic and mediastinal disorders) | 42 | 19
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 22 | 6
Decreased appetite (Metabolism and nutrition disorders) | 28 | 18
Insomnia (Psychiatric disorders) | 23 | 13
Dyspepsia (Gastrointestinal disorders) | 19 | 14
Lymphocyte count decreased (Investigations) | 53 | 20
Platelet count decreased (Investigations) | 19 | 11
Hypokalaemia (Metabolism and nutrition disorders) | 19 | 5
Back pain (Musculoskeletal and connective tissue disorders) | 18 | 11

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.